CLINICAL TRIAL: NCT01988506
Title: Induction of Regulatory t Cells by Low Dose IL2 in Autoimmune and Inflammatory Diseases: a Transnosographic Approach
Brief Title: Induction of Regulatory t Cells by Low Dose il2 in Autoimmune and Inflammatory Diseases
Acronym: TRANSREG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130101; 2013-001232-22 (EudraCT Number)
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Systemic Lupus Erythematosus; Psoriasis; Behcet's Disease; Wegener's Granulomatosis; Takayasu's Disease; Crohn's Disease; Ulcerative Colitis; Autoimmune Hepatitis; Sclerosing Cholangitis; Gougerot-sjögren; Idiopathic Thrombocytopenic Purpura; Systemic Sclerosis
Keywords: IL2,; Interleukin 2,; ILT101; Proleukin®, RhIL-2; Auto-immune disease; Inflammatory disease; Inflammation; Regulatory T cells,; Treg; Immunoregulation; Immune tolerance
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Lupus Erythematosus, Systemic; Psoriasis; Behcet Syndrome; Granulomatosis with Polyangiitis; Aortic Arch Syndromes; Crohn Disease; Colitis, Ulcerative; Hepatitis, Autoimmune; Cholangitis, Sclerosing; Purpura, Thrombocytopenic, Idiopathic; Scleroderma, Systemic; Inflammation | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interleukin 2 (Experimental): Interleukin 2, 1MUI.= Proleukin®, RhIL-2
  Interventions: Drug: Interleukin 2

INTERVENTIONS:
Drug: Interleukin 2 — Induction period: repeated administration of low-dose IL-2 (1MUI/day, sc) during 5 consecutive days.Maintenance period: treatment with IL-2, 1MUI once every 15 days (except systemic lupus erythematosus's patients every 7 days) for 6 months

SUMMARY:
TRANSREG will assess the safety and biological efficacy of low-dose IL2 as a Treg inducer in a set of 14 autoimmune and auto-inflammatory diseases, with the aim to select diseases in which further therapeutic development will be performed. Extensive biological- and immune-monitoring pre- and post-IL2 will contribute (i) to define the common or distinct processes responsible for the breakdown of immunological tolerance in these pathologies and (ii) to discover potential biomarkers of the IL2 response.

DETAILED DESCRIPTION:
Protocol: TRANSREG is a multicentric, uncontrolled, open-label study, comparing biological and clinical responses to the administration of low doses IL2 across 14 selected pathologies: rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, psoriasis, Behcet's disease, Wegener's granulomatosis, Takayasu's disease, Crohn's disease, ulcerative colitis, autoimmune hepatitis, sclerosing cholangitis, Gougerot-sjögren, Systemic Sclerosis and Idiopathic Thrombocytopenic Purpura. Methods: Each patient will receive 1MUI /day of IL2 from Day-1 to Day-5 (the induction period), and then every 2 weeks (except systemic lupus erythematosus's patients will received every week) from Day-15 to Day-180 (the maintenance period). Patients will thereafter be followed up for 12 months (Day-181-Day-540). For each pathology, 6 patients will be included at Pitié-Salpêtrière, Cochin, Saint Antoine, Paul Brousse and Henri Mondor hospitals in Paris and Créteil, France. An interim analysis will be performed in each pathology group when the first six patients have received at least 3 months of treatment. In those pathology groups in which a Treg response will be documented, six additional patients will be included. In total, a minimum of 84 patients and up to 132 patients will be enrolled in this study. Primary efficacy endpoint is the Treg response at Day-8 compared to baseline. Secondary efficacy endpoints are:- evolution of the Treg response during the maintenance period,- the changes in markers of inflammation - the clinical response, evaluated by means of global generic scales [Clinical Global Impression severity scale (CGI-sev) and Clinical Global Impression efficacy index (CGI-eff)] as well as specific clinical and biological evaluations for each disease, - the frequency of relapses, - the assessment of quality of life (scale EuroQL-5). Expected Results: TRANSREG will define which patients respond to IL2, whether per pathology or according to pre-treatment phenomics, allowing to guide further clinical development of low dose IL2 in autoimmune and auto-inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 year
* male or female
* documented diagnosis of one AIID among the 14 diseases selected (following consensual specific criteria)
* stable or moderately active disease (except Lupus) under standard treatment (≥ 2 months) at the time of inclusion (except Sclerosing Cholangitis, Gougerot-sjögren, Takayasu's Disease and Systemic Sclerosis)
* normal thyroid function (with or without treatment)
* effective contraception for more than two weeks at inclusion and negative beta HCG test for women of childbearing potential,
* affiliated to the social security system
* written informed consent form.

Exclusion Criteria:

* known intolerance for IL2 (see SPC),
* administration of a non-authorized treatment and/or IV bolus of corticosteroids in the last 2 months,
* vaccination with live attenuated virus in the months preceding the inclusion or planned during the study
* other severe or progressive autoimmune/inflammatory pathology,
* low white blood cell count<2000/mm3, lymphocytes <600/mm3, platelets <80 000/mm3,
* heart failure (≥ grade III NYHA), renal insufficiency (Cockcroft< 60ml/mn except patients with lupus or Wegener's granulomatosis) or hepatic insufficiency (transaminases> 5N except for patients with autoimmune hepatitis), or lung failure,
* significant abnormality in chest X-ray other than these linked to the diseases under investigation
* cancer or history of cancer cured for less than five years (except in situ carcinoma of the cervix or basocellular carcinoma)
* poor venous access not allowing repeated blood tests,
* restrictive diet or parenteral nutrition,
* surgery during the last 2 months or surgery planned during the study,
* participation in other biomedical research in the last 3 months or planned during the study.
* pregnant or lactating women,
* concomitant psychiatric disease or any other chronic illness or drug-abuse that could interfere with the ability to comply with the protocol or to give informed consent,
* positive HIV serology, active hepatitis B or EBV infection,
* patients under a measure of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Percentages of Tregs | Day8
  Change in Treg percentage (percentages of Tregs within the CD4+ lymphocytes) at Day-8 after administration of low-dose of IL2 compared to baseline (Day0)

SECONDARY OUTCOMES:
Percentages of Tregs | Day 15, 29, 85, 183, 240, 360 and 540
  Changes in Treg percentage at Day 15, 29, 85, 183, 240, 360 and 540 compared to baseline (Day0)
inflammation markers (CRP and CRP ultra sensible) | Day 0, 1, 8, 15, 29, 85, 183, 240, 360 and 540
  Changes in levels of inflammation markers
markers of inflammatory anemia (Hemoglobin, serum iron level, transferrin) ferritin | Day 0, 1, 8, 15, 29, 85, 183, 240, 360 and 540
  Changes in levels of inflammation markers
Number of relapses | up to Day540
CGI-sev, CGI-activity and CGI-eff scales | Day 85, 183, 240, 360 and 540
  Change in the clinical global impression severity and efficacy scale (CGI-sev, CGI-act and CGI-eff scales) at Day 85, 183, 240, 360 and 540 compared to baseline (Day1)
EuroQL-5 scale | Day 183
  Change in the quality of life (EuroQL-5 scale)
Evolution of clinical, biological or radiological criteria specific to each disease | up to Day 540
  Changes in disease-specific score and/or evolution of clinical, biological or radiological criteria specific to each disease
Safety Assessment | up to Day 540
  Safety Assessment all along the observation period (Day-1 to Day-240): Safety assessment will include vital signs, adverse events and concomitant medications collection as well as biology during the 6 months of the treatment period; .In addition, the evolution of the disease will be followed up to 1 year after IL2- treatment stop.

CONTACTS AND LOCATIONS:
Overall Officials: David KLATZMANN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (11):
- France (11):
  - Henri Mondor - Médecine Interne, Créteil
  - Médecine interne - Hôpital Saint-Antoine, Paris
  - Service de médecine vasculaire - HEGP, Paris
  - Service d' Hépato Gastro Entérologie - Hôpital SAINT-ANTOINE, Paris, Île-de-France Region
  - Service de Gastro Entérologie - Hôpital SAINT-ANTOINE, Paris, Île-de-France Region
  - Service de Rhumatologie - Hôpital SAINT-ANTOINE, Paris, Île-de-France Region
  - CIC - Hôpital PITIE SALPETRIERE, Paris, Île-de-France Region
  - Service de Médecine Interne - Hôpital PITIE SALPETRIERE, Paris, Île-de-France Region
  - Service de Rhumatologie - Hôpital PITIE SALPETRIERE, Paris, Île-de-France Region
  - Service de Dermatologie - Hôpital COCHIN, Paris, Île-de-France Region
  - Centre Hépato-Biliaire - Hôpital Paul Brousse, Villejuif, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenzwajg M, Lorenzon R, Cacoub P, Pham HP, Pitoiset F, El Soufi K, RIbet C, Bernard C, Aractingi S, Banneville B, Beaugerie L, Berenbaum F, Champey J, Chazouilleres O, Corpechot C, Fautrel B, Mekinian A, Regnier E, Saadoun D, Salem JE, Sellam J, Seksik P, Daguenel-Nguyen A, Doppler V, Mariau J, Vicaut E, Klatzmann D. Immunological and clinical effects of low-dose interleukin-2 across 11 autoimmune diseases in a single, open clinical trial. Ann Rheum Dis. 2019 Feb;78(2):209-217. doi: 10.1136/annrheumdis-2018-214229. Epub 2018 Nov 24. PMID 30472651